CLINICAL TRIAL: NCT04881838
Title: Using a Modified ALCL99 Regimen for Chinese Children with Newly Diagnosed High-risk Anapestic Large Cell Lymphoma
Brief Title: CCCG-ALCL-2020 for Chinese Children and Adolescents with Newly Diagnosed High-risk ALCL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Cancer Group, China (Network)
Collaborators: Shanghai Children's Medical Center (Other); Nanjing Children's Hospital (Other); Qilu Hospital of Shandong University (Other); Tianjin Cancer Hospital (Unknown); West China Second University Hospital (Other); Xiangya Hospital (Other); 1st Affiliated Hospital of Zhengzhou University (Unknown); Shenzhen Children's Hospital (Other Government); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCCG-ALCL-2020
Record Dates: First submitted 2021-05-10; First posted 2021-05-11 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Pediatric Anaplastic Large Cell Lymphoma
Keywords: Anapestic Large Cell Lymphoma; vinorelbine; pediatric; treatment outcome; Chinese
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic | interventions — Maintenance

STUDY DESIGN:
Intervention Model Description: All enrolled patients stratified into high risk group are assigned to one treatment regimen
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- High risk group (Experimental): 1. Stage I, unresected; Stage I with "B" syndrome
  2. Stage II
  3. Stage III
  4. Stage IV without CNS involvement
  Interventions: Drug: P regimen; Drug: Course A1 + Vin; Drug: Course B1 +Vin; Drug: Course A2 + Vin; Drug: Course B2 +Vin; Drug: Course A3 + Vin; Drug: Course B3 +Vin; Drug: Maintenance therapy

INTERVENTIONS:
Drug: P regimen — Dexamethasone 5 mg/m2 Days 1 and 2; 10mg/m2 Day 3 to 5; Cyclophosphamide 200 mg/m2 Days 1 and 2 Intrathecal therapy Day 1
Drug: Course A1 + Vin — vinorelbine 25 mg/m2, Day 1 Dexamethasone 10 mg/m2 Days 1 to 5; Methotrexate 3g/m2, 3-hour infusion Day 1; Etoposide 100mg/m2, Days 4 to 5; Ifosfamide 800 mg/m2, Days 1 to 5; Cytarabine 150 mg/m2, q12h Days 4 to 5;
Drug: Course B1 +Vin — vinorelbine 25 mg/m2, Day 1; Dexamethasone 10 mg/m2 Days 1 to 5; Methotrexate 3g/m2, 3-hour infusion Day 1; Cyclophosphamide 200 mg/m2, Days 1 to 5; Doxorubicin 25 mg/m2, Days 4 to 5;
Drug: Course A2 + Vin — vinorelbine 25 mg/m2, Day 1 Dexamethasone 10 mg/m2 Days 1 to 5; Methotrexate 3g/m2, 3-hour infusion Day 1; Etoposide 100mg/m2, Days 4 to 5; Ifosfamide 800 mg/m2, Days 1 to 5; Cytarabine 150 mg/m2, q12h Days 4 to 5;
Drug: Course B2 +Vin — vinorelbine 25 mg/m2, Day 1; Dexamethasone 10 mg/m2 Days 1 to 5; Methotrexate 3g/m2, 3-hour infusion Day 1; Cyclophosphamide 200 mg/m2, Days 1 to 5; Doxorubicin 25 mg/m2, Days 4 to 5;
Drug: Course A3 + Vin — vinorelbine 25 mg/m2, Day 1 Dexamethasone 10 mg/m2 Days 1 to 5; Methotrexate 3g/m2, 3-hour infusion Day 1; Etoposide 100mg/m2, Days 4 to 5; Ifosfamide 800 mg/m2, Days 1 to 5; Cytarabine 150 mg/m2, q12h Days 4 to 5;
Drug: Course B3 +Vin — vinorelbine 25 mg/m2, Day 1; Dexamethasone 10 mg/m2 Days 1 to 5; Methotrexate 3g/m2, 3-hour infusion Day 1; Cyclophosphamide 200 mg/m2, Days 1 to 5; Doxorubicin 25 mg/m2, Days 4 to 5;
Drug: Maintenance therapy — Vinorelbine 25 mg/m2 IV, weekly for 3 consecutive weeks followed by 1-week rest. Totally 80 cycles.

SUMMARY:
A prospective study on the efficacy of modified ALCL99 regimens in the treatment of the current Chinese pediatric and adolescent high-risk ALCL and compared with our historical data.

DETAILED DESCRIPTION:
Anaplastic large cell lymphoma (ALCL) accounts for 15% of pediatric and adolescent non-Hodgkin lymphomas (NHLs). In our historical study (retrospective multicenter study), the 3-year event-free survival (EFS) was 65% for 80 eligible patients treated in 10 centers between January 2009 and June 2014.

The ALCL99 trial reported a 2-year overall survival of 92% and 2-year event-free survival of 74% then become the current standard frontline treatment for pediatric ALCL. The recent long-term follow-up data from ALCL99 trial highlighted its excellent outcome. A less toxic schedule of methotrexate (MTX) 3g/m2 in a 3-hour infusion without intrathecal therapy reproduced the favorable results from previous reports of NHL-BFM90 protocol with MTX at 1g/m2 in a 3-hour infusion. Additionally, a prospective ALCL-Relapse trial by the European Inter-Group for Childhood Non-Hodgkin Lymphoma demonstrated 80% of patients with a late relapse can be cured by 24 months of vinblastine monotherapy. However, vinblastine would not be advised as a treatment option in mainland China due to its inaccessibility. A pilot experience using single-drug vinorelbine in 4 pediatric patients with relapsed ALCL with satisfactory outcome provides the rational for studying vinorelbine as a front line drug option.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be ≤ 18 years at the time of diagnosis
* Newly diagnosed patients with histologically confirmed high-risk anaplastic large cell lymphoma
* No congenital immunodeficiency, HIV infection, or prior organ transplant

Exclusion Criteria:

* Patients have received prior cytotoxic chemotherapy/target therapy/radiation, if any steroid applied, total prior steroids dosage > Dexamethasone 40 mg/m2 for the current diagnosis or any cancer
* Patients have overwhelming infection, and a life expectancy of < 2 weeks

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 172 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
3-year event free survival (EFS) | Up to 3 years
  Calculated from the time of diagnosis to the first of the following events: progression, relapse, secondary ,malignancy or death
Treatment-related adverse events | Up to 3years
  Number of participants with treatment-related adverse events as assessed by CTCAEv5.0

SECONDARY OUTCOMES:
Patient compliance | Up to 3years
  the percentage of patients who complete the maintenance therapy of this modified ALCL99 regimens
Value of early PET/CT in pediatric ALCL | Up to 3 years
  Prognostic value of early remission of PET/CT after 2 cycles of chemotherapy in pediatric ALCL
Value of peripheral blood or bone marrow NPM-ALK or ALK-variants level in pediatric ALCL | Up to 3 years
  Prognostic value of peripheral blood/bone marrow NPM-ALK or ALK-variants level (qPCR) at diagnosis in pediatric ALCL

CONTACTS AND LOCATIONS:
Overall Officials: Yijin Gao, MD, Principal Investigator — Shanghai Children's Medical Center
Locations (1):
- Shanghai Children's Medical Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, SAP and ICF were shared before study initiation. Patient data and the information about the process of the study will be shared within the all participants annually after enrollment patients.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be shared within the all hospitals every 12 months after enrollment of patients.
Access Criteria: Scheduled meeting and paper transferring.

REFERENCES:
- [Background] Mussolin L, Le Deley MC, Carraro E, Damm-Welk C, Attarbaschi A, Williams D, Burke A, Horibe K, Nakazawa A, Wrobel G, Mann G, Csoka M, Uyttebroeck A, Fernandez-Delgado Cerda RF, Beishuizen A, Mellgren K, Burkhardt B, Klapper W, Turner SD, D'Amore ESG, Lamant L, Reiter A, Woessmann W, Brugieres L, Pillon MPOBOTEIFCNL. Prognostic Factors in Childhood Anaplastic Large Cell Lymphoma: Long Term Results of the International ALCL99 Trial. Cancers (Basel). 2020 Sep 24;12(10):2747. doi: 10.3390/cancers12102747. PMID 32987765
- [Background] Knorr F, Brugieres L, Pillon M, Zimmermann M, Ruf S, Attarbaschi A, Mellgren K, Burke GAA, Uyttebroeck A, Wrobel G, Beishuizen A, Aladjidi N, Reiter A, Woessmann W; European Inter-Group for Childhood Non-Hodgkin Lymphoma. Stem Cell Transplantation and Vinblastine Monotherapy for Relapsed Pediatric Anaplastic Large Cell Lymphoma: Results of the International, Prospective ALCL-Relapse Trial. J Clin Oncol. 2020 Dec 1;38(34):3999-4009. doi: 10.1200/JCO.20.00157. Epub 2020 Jul 30. PMID 32730187
- [Background] Yuan Q, He Q, Mi Q, Yin MZ, Han YL, Gao YJ. Single-drug vinorelbine as a salvage re-induction regimen for 4 consecutive pediatric patients with relapsed anaplastic large-cell lymphoma in a single children's institution. Ann Hematol. 2021 Apr;100(4):1093-1095. doi: 10.1007/s00277-020-04175-3. Epub 2020 Jul 13. No abstract available. PMID 32661576
- [Background] Le Deley MC, Rosolen A, Williams DM, Horibe K, Wrobel G, Attarbaschi A, Zsiros J, Uyttebroeck A, Marky IM, Lamant L, Woessmann W, Pillon M, Hobson R, Mauguen A, Reiter A, Brugieres L. Vinblastine in children and adolescents with high-risk anaplastic large-cell lymphoma: results of the randomized ALCL99-vinblastine trial. J Clin Oncol. 2010 Sep 1;28(25):3987-93. doi: 10.1200/JCO.2010.28.5999. Epub 2010 Aug 2. PMID 20679620
- [Background] Brugieres L, Le Deley MC, Rosolen A, Williams D, Horibe K, Wrobel G, Mann G, Zsiros J, Uyttebroeck A, Marky I, Lamant L, Reiter A. Impact of the methotrexate administration dose on the need for intrathecal treatment in children and adolescents with anaplastic large-cell lymphoma: results of a randomized trial of the EICNHL Group. J Clin Oncol. 2009 Feb 20;27(6):897-903. doi: 10.1200/JCO.2008.18.1487. Epub 2009 Jan 12. PMID 19139435
- [Background] Lymphoma Study Group, Subspecialty Group of Hematology, the Society of Pediatrics, Chinese Medical Association; Lymphoma Study Group, Committee of Pediatrics, Chinese Anti-Cancer Association. [Diagnosis and treatment of anaplastic large-cell lymphoma in children and adolescents: a retrospective multicenter survey study]. Zhonghua Er Ke Za Zhi. 2017 Mar 2;55(3):194-199. doi: 10.3760/cma.j.issn.0578-1310.2017.03.006. Chinese. PMID 28273702
- [Background] Mosse YP, Voss SD, Lim MS, Rolland D, Minard CG, Fox E, Adamson P, Wilner K, Blaney SM, Weigel BJ. Targeting ALK With Crizotinib in Pediatric Anaplastic Large Cell Lymphoma and Inflammatory Myofibroblastic Tumor: A Children's Oncology Group Study. J Clin Oncol. 2017 Oct 1;35(28):3215-3221. doi: 10.1200/JCO.2017.73.4830. Epub 2017 Aug 8. PMID 28787259